CLINICAL TRIAL: NCT03957850
Title: Cognitive Reappraisal in Adolescents With Major Depression: From Neurobiological Mechanisms to Intervention
Brief Title: Cognitive Reappraisal in Adolescents With Major Depression
Acronym: KONNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Research Foundation (Other); RWTH Aachen University (Other); University of Amsterdam (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Postdoctoral Researcher, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 399482529
Record Dates: First submitted 2019-05-03; First posted 2019-05-21 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder
Keywords: Emotion Regulation Training; LPP; Adolescence; Major Depression; Eye-tracking; Cognitive Reappraisal; Event-related Potentials
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This study is designed as a short-term randomized controlled, participant-blind clinical trial including two groups of adolescents with MD. MD participants will be randomly assigned to a group that receives task-based training in CR or to a control training. Randomisation will be performed by a statistician, stratifying for age (14 years and younger and 15 years and older) and sex.
Who Masked: Participant
Masking Description: Participant-blind clinical trial: the participants are blinded regarding the allocation to the respective training group (CR training or control training). Upon completion of the training (including questionnaire assessment), participants are unblinded regarding the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Reappraisal Training Group (Experimental): Cognitive Reappraisal Training group will perform 4 training sessions in Cognitive Reappraisal during which, behavioral responses, event-related potentials (ERPs) and eye-tracking data are collected.
  Interventions: Behavioral: Cognitive Reappraisal Training
- Control Training Group (Active Comparator): Control Training Group will perform 4 control sessions without Cognitive Reappraisal Training during which behavioral responses, ERP and eye-tracking data are collected.
  Interventions: Behavioral: Control Training

INTERVENTIONS:
Behavioral: Cognitive Reappraisal Training — The training procedure is adapted from a study by Denny & Ochsner (2014). Before the task, participants are instructed that they will be presented pictures and that these pictures will be preceded by a condition specific cue signaling the appropriate strategy during picture viewing. Participants are instructed to indicate their affective response to the image on a rating scale. The task involves 4 conditions: 1) Negative-decrease: participants are asked to view negative pictures and to decrease their affective response by reappraising the negative event. 2) Negative-attend/ 3) Neutral-attend/ 4) Positive-attend: participants are asked to view pictures and to respond naturally to them without trying to alter their affective response. The training task will be repeated over 4 training sessions.
  Arms: Cognitive Reappraisal Training Group
Behavioral: Control Training — The task in the control group is implemented to account for unspecific effects and is as similar as possible to the CR task except that it involves no negative-decrease (i.e., no reappraisal) condition. Instead, the control task only involves the three attend conditions (negative- attend, neutral-attend, positive-attend).
  Arms: Control Training Group

SUMMARY:
Major depression (MD) is common during adolescence and associated with significant morbidity and mortality. One important factor for the development and maintenance of adolescent MD are disturbances in emotion regulation, including deficits in cognitive reappraisal (CR). CR is a particularly effective emotion regulation strategy that aims at reinterpreting emotional events to modify affective responses. Adolescents with MD apply this strategy less often than their healthy peers and show disturbances in brain activation patterns underlying CR.

In this study, MD adolescents will be randomly assigned to a group that receives a task-based training in CR or to a control training group. It will be examined whether the task-based CR training is superior to the control training with regard to improvements in negative affect, perceived stress in daily life and depressive symptoms. Moreover, during the four training sessions, the event-related potential "Late Positive Potential" (LPP) will be recorded to assess neurophysiological indices of CR processes and gaze fixations on emotional areas within negative pictures and affective responses to pictures will be collected to identify mechanisms underlying training effects.This study will provide first evidence for the efficacy of a short-time training that has previously shown to be effective in healthy individuals. Moreover, the study will identify neurobiological mechanisms that predict training effects. The results of this investigation will lay the ground for a clinical trial to investigate whether a CR training added to an established intervention improves treatment effects for adolescent MD.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants
* age range: 12-18 years
* current diagnosis of MD (ICD-10 diagnoses F32.0; F32.1; F32.2, F33.0, F33.1, F.33.2)
* intelligence quotient (IQ) of ≥ 80

Exclusion Criteria:

* neurological disorders
* schizophrenic disorder
* pervasive developmental disorder
* bipolar disorder
* borderline personality disorder
* substance dependence disorder
* gender dysphoria.

Participants comorbid with psychiatric comorbidities other than those listed above are included if MD is the primary diagnosis.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Change in negative and positive affect via the Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | Over the course of the four training sessions, which will take place within the time frame of two weeks. This outcome measure will be reassessed at follow-up (2 weeks after the end of the entire training).
  A change in negative affect will be assessed based on the Negative Affect scale of the PANAS-C-SF. This scale ranges from one to five, with higher scores indicating more negative affect. A change in positive affect will be assessed based on the Positive Affect scale of the PANAS-C-SF. This scale ranges from one to five, with higher scores indicating more positive affect.
Change in perceived stress via the Perceived Stress Scale (PSS-10) | During each of the four training sessions, which will take place within the time frame of two weeks. This outcome measure will be reassessed at follow-up (two weeks after the end of the training sessions).
  Change in perceived stress will be assessed based on the German adaption of the PSS-10. This scale ranges from 1-5, with higher scores indicating more perceived stress.
Change in rumination as assessed via the German adaptation of the Response Style Questionnaire (RSQ-D) | Pretraining & after completion of the last of four training session. The training sessions will take place within the time frame of two weeks. This outcome measure will be reassessed at follow-up (two weeks after the end of the training sessions).
  Change in rumination will be assessed based on two separate rumination subscales of the RSQ-D. The self-focused rumination scale ranges from 7-28, with higher scores indicating higher self-focused rumination. The symptom-focused rumination scale ranges from 8-31, with higher scores indicating higher symptom-focused rumination.
Change in depressive Symptoms via the Beck Depression Inventory - Second Edition (BDI-II) | Pretraining & after completion of the last of four training session. The training sessions will take place within the time frame of two weeks.
  Change in depressive symptoms will be assessed based on the BDI-II. This scale ranges from 0-63, with higher scores indicated more depressive symptoms.

SECONDARY OUTCOMES:
Changes in the downregulation of affective behavioral responses to negative pictures via CR based on the self-assessment manikin scale | During each of the four training sessions, which will take place within the time frame of two weeks.
  Affective behavioral responses to negative pictures will be continuously assessed during each of the four training sessions. This assessment is based on the self-assessment manikin scale for valence (Bradley & Lang, 1994), which is a 9-point rating scale with higher scores indicating higher positive affect. To obtain a behavioral index of downregulated affect in the CR training group, averaged behavioral affective responses during an attend condition will be subtracted from averaged behavioral affective responses during an active regulate condition.
Changes in the downregulation of the LPP (late positive potential) to negative pictures via CR | During each of the four training sessions, which will take place within the time frame of two weeks.
  The LPP elicited to negative pictures will be continuously assessed during each of the four training sessions. To calculate the downregulation of the LPP via CR in the CR training group, the averaged LPP during an attend condition will be subtracted from the averaged LPP during an active regulate condition.
Changes in the percent gaze fixations in emotional areas of interest within negative pictures | During each of the four training sessions, which will take place within the time frame of two weeks.
  Changes in the percent duration of gaze fixations within a-priori defined emotional interest areas within negative pictures will be exploratively assessed over the course of the four training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Greimel, PhD, Principal Investigator — Department of Child&Adolescent Psychiatry, Psychosomatics&Psychoth.,LMU Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich, Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data in our study contains sensitive patient information, such as sociodemographic information and comorbidities. Since patients could possibly be identified by making our raw data publicly available, ethical principles of protecting patient confidentiality would be breached. Aggregated group data can be made available upon request.

REFERENCES:
- [Background] Denny BT, Ochsner KN. Behavioral effects of longitudinal training in cognitive reappraisal. Emotion. 2014 Apr;14(2):425-33. doi: 10.1037/a0035276. Epub 2013 Dec 23. PMID 24364856
- [Background] Bradley MM, Lang PJ. Measuring emotion: the Self-Assessment Manikin and the Semantic Differential. J Behav Ther Exp Psychiatry. 1994 Mar;25(1):49-59. doi: 10.1016/0005-7916(94)90063-9. PMID 7962581
- [Derived] Zsigo C, Feldmann L, Oort F, Piechaczek C, Bartling J, Schulte-Ruther M, Wachinger C, Schulte-Korne G, Greimel E. Emotion regulation training for adolescents with major depression: Results from a randomized controlled trial. Emotion. 2024 Jun;24(4):975-991. doi: 10.1037/emo0001328. Epub 2023 Dec 7. PMID 38060020
- [Derived] Greimel E, Feldmann L, Piechaczek C, Oort F, Bartling J, Schulte-Ruther M, Schulte-Korne G. Study protocol for a randomised-controlled study on emotion regulation training for adolescents with major depression: the KONNI study. BMJ Open. 2020 Sep 10;10(9):e036093. doi: 10.1136/bmjopen-2019-036093. PMID 32912977